CLINICAL TRIAL: NCT04760756
Title: The Effects of Fragility Fracture Integrated Rehabilitation Management (FIRM) of Hip Fracture in Geriatrics
Brief Title: The Effects of Fragility Fracture Integrated Rehabilitation Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zohra Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Aftab, Assistant Professor, Zohra Institute of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/0045 Anam Aftab
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-08

CONDITIONS: Hip Fractures
Keywords: Activities of daily living; Mobility limitation; Occupational Therapy; Physical Therapy
MeSH Terms: conditions — Hip Fractures; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This refers to Fragility Fracture Integrated Rehabilitation Management (Experimental): This refers to Fragility Fracture Integrated Rehabilitation Management and will include comprehensive rehabilitation program and assessment
  Interventions: Other: Fragility Fracture Integrated Rehabilitation Management

INTERVENTIONS:
Other: Fragility Fracture Integrated Rehabilitation Management — * At least 2 hours of rehabilitation management per day
  * Including occupational therapy (training to improve daily life performance)
  * Inpatient (the first 2 weeks): daily management (body control ability, mobility ability, hygiene management, etc.)
  * Outpatient (2-6 weeks): management once a week
  * The management period is for 2 weeks (1 week after surgery)

SUMMARY:
• To determine the effects of Fragility Fracture Integrated Rehabilitation Management approach in geriatric hip fracture patients (post surgical)

DETAILED DESCRIPTION:
This refers to Fragility Fracture Integrated Rehabilitation Management and will include following comprehensive rehabilitation program including rehab specialist, physiotherapist, occupational therapist and rehab nurse.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above 55 years of age, who underwent hip fracture management NIRM Pakistan due to hip fracture
2. Patient diagnosed with femur neck, intertrochanteric fracture, and sub-trochanteric fracture
3. Patient who got bipolar hemiarthroplasty, total hip replacement arthroplasty, reduction and internal fixation

Exclusion Criteria:

1. Patients who underwent surgery for a cause other than a hip fracture (infection, arthritis, loosening, avascular necrosis)
2. Patients who underwent surgery because of femur shaft fracture, acetabular fracture, periprosthetic fracture pathologic fracture by tumor
3. Isolated fracture of the greater or lesser tuberosity
4. Multiple fracture
5. Revision operation
6. Patients who do not agree to participate in clinical trials

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Functional Ambulatory Category (FAC) | 2 weeks
  The Functional Ambulation Categories (FAC) is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device
EQ-5D | 2 weeks
  EQ-5D is a standardized instrument for measuring generic health status. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Modified Barthel index (MBI) | 2 weeks
  Modified Barthel ADL index Measure of physical disability used widely to assess behaviour relating to activities of daily living for patients with disabling conditions. It measures what patients do in practice.

CONTACTS AND LOCATIONS:
Overall Officials: Anam Aftab, Phd*, Principal Investigator — Riphah college of rehabilitation and allied health sciences - Rawalpindi
Locations (1):
- National Institute of Rehabilitation Medicine, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boschitsch EP, Durchschlag E, Dimai HP. Age-related prevalence of osteoporosis and fragility fractures: real-world data from an Austrian Menopause and Osteoporosis Clinic. Climacteric. 2017 Apr;20(2):157-163. doi: 10.1080/13697137.2017.1282452. Epub 2017 Feb 8. PMID 28286986
- [Background] Nanes MS, Kallen CB. Clinical assessment of fracture risk and novel therapeutic strategies to combat osteoporosis. Fertil Steril. 2009 Aug;92(2):403-12. doi: 10.1016/j.fertnstert.2009.05.049. Epub 2009 Jun 25. PMID 19559412
- [Background] Kanis JA, Melton LJ 3rd, Christiansen C, Johnston CC, Khaltaev N. The diagnosis of osteoporosis. J Bone Miner Res. 1994 Aug;9(8):1137-41. doi: 10.1002/jbmr.5650090802. No abstract available. PMID 7976495
- [Background] Watts NB, Bilezikian JP, Camacho PM, Greenspan SL, Harris ST, Hodgson SF, Kleerekoper M, Luckey MM, McClung MR, Pollack RP, Petak SM; AACE Osteoporosis Task Force. American Association of Clinical Endocrinologists Medical Guidelines for Clinical Practice for the diagnosis and treatment of postmenopausal osteoporosis. Endocr Pract. 2010 Nov-Dec;16 Suppl 3(Suppl 3):1-37. doi: 10.4158/ep.16.s3.1. No abstract available. PMID 21224201
- [Background] Devereux G, Litonjua AA, Turner SW, Craig LC, McNeill G, Martindale S, Helms PJ, Seaton A, Weiss ST. Maternal vitamin D intake during pregnancy and early childhood wheezing. Am J Clin Nutr. 2007 Mar;85(3):853-9. doi: 10.1093/ajcn/85.3.853. PMID 17344509
- [Background] Khan K, Brown J, Way S, Vass N, Crichton K, Alexander R, Baxter A, Butler M, Wark J. Overuse injuries in classical ballet. Sports Med. 1995 May;19(5):341-57. doi: 10.2165/00007256-199519050-00004. PMID 7618011
- [Background] Shane E, Burr D, Ebeling PR, Abrahamsen B, Adler RA, Brown TD, Cheung AM, Cosman F, Curtis JR, Dell R, Dempster D, Einhorn TA, Genant HK, Geusens P, Klaushofer K, Koval K, Lane JM, McKiernan F, McKinney R, Ng A, Nieves J, O'Keefe R, Papapoulos S, Sen HT, van der Meulen MC, Weinstein RS, Whyte M; American Society for Bone and Mineral Research. Atypical subtrochanteric and diaphyseal femoral fractures: report of a task force of the American Society for Bone and Mineral Research. J Bone Miner Res. 2010 Nov;25(11):2267-94. doi: 10.1002/jbmr.253. PMID 20842676
- [Background] Holroyd C, Cooper C, Dennison E. Epidemiology of osteoporosis. Best Pract Res Clin Endocrinol Metab. 2008 Oct;22(5):671-85. doi: 10.1016/j.beem.2008.06.001. PMID 19028351
- [Background] Shepstone L, Fordham R, Lenaghan E, Harvey I, Cooper C, Gittoes N, Heawood A, Peters T, O'Neill T, Torgerson D, Holland R, Howe A, Marshall T, Kanis J, McCloskey E. A pragmatic randomised controlled trial of the effectiveness and cost-effectiveness of screening older women for the prevention of fractures: rationale, design and methods for the SCOOP study. Osteoporos Int. 2012 Oct;23(10):2507-15. doi: 10.1007/s00198-011-1876-7. PMID 22314936
- [Background] Kanis JA, Johnell O, Oden A, Johansson H, McCloskey E. FRAX and the assessment of fracture probability in men and women from the UK. Osteoporos Int. 2008 Apr;19(4):385-97. doi: 10.1007/s00198-007-0543-5. Epub 2008 Feb 22. PMID 18292978
- [Background] Cummings SR, Kelsey JL, Nevitt MC, O'Dowd KJ. Epidemiology of osteoporosis and osteoporotic fractures. Epidemiol Rev. 1985;7:178-208. doi: 10.1093/oxfordjournals.epirev.a036281. No abstract available. PMID 3902494
- [Background] Riggs BL, Melton LJ 3rd. The worldwide problem of osteoporosis: insights afforded by epidemiology. Bone. 1995 Nov;17(5 Suppl):505S-511S. doi: 10.1016/8756-3282(95)00258-4. PMID 8573428
- [Background] Bukata SV, Digiovanni BF, Friedman SM, Hoyen H, Kates A, Kates SL, Mears SC, Mendelson DA, Serna FH Jr, Sieber FE, Tyler WK. A guide to improving the care of patients with fragility fractures. Geriatr Orthop Surg Rehabil. 2011 Jan;2(1):5-37. doi: 10.1177/2151458510397504. No abstract available. PMID 23569668
- [Background] Coleman EA. Falling through the cracks: challenges and opportunities for improving transitional care for persons with continuous complex care needs. J Am Geriatr Soc. 2003 Apr;51(4):549-55. doi: 10.1046/j.1532-5415.2003.51185.x. PMID 12657078
- [Background] Kates SL, Mendelson DA, Friedman SM. Co-managed care for fragility hip fractures (Rochester model). Osteoporos Int. 2010 Dec;21(Suppl 4):S621-5. doi: 10.1007/s00198-010-1417-9. Epub 2010 Nov 6. PMID 21058002
- [Background] Thompson PD, Buchner D, Pina IL, Balady GJ, Williams MA, Marcus BH, Berra K, Blair SN, Costa F, Franklin B, Fletcher GF, Gordon NF, Pate RR, Rodriguez BL, Yancey AK, Wenger NK; American Heart Association Council on Clinical Cardiology Subcommittee on Exercise, Rehabilitation, and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism Subcommittee on Physical Activity. Exercise and physical activity in the prevention and treatment of atherosclerotic cardiovascular disease: a statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity). Circulation. 2003 Jun 24;107(24):3109-16. doi: 10.1161/01.CIR.0000075572.40158.77. No abstract available. PMID 12821592